CLINICAL TRIAL: NCT02056873
Title: The Human Thalamocortical Network in Tourette Syndrome
Brief Title: Tourette Syndrome Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Medtronic (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201300850 -A-N; R01NS096008 (NIH); 1553482 (Other Grant/Funding Number: NATIONAL SCIENCE FOUNDATION); OCR20343 (Other: UF OnCore)
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Tourette Syndrome
Keywords: deep brain stimulation; DBS; tourette; tourette's; tourette syndrome; TS
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Deep Brain Stimulation (DBS) (Experimental): Subjects' DBS surgical intervention requires implantation of a DBS system: two CM thalamic leads (one in each brain hemisphere), two ECOG strip leads (one in each brain hemisphere), and two neurostimulators implanted in the chest.
  The ECOG strip lead is implanted into the brain to provide an interface through which stimulation can be delivered or activity of the brain can be monitored by the device, or observed by a clinician using a programmer.
  Neurostimulator and leads system includes a programmer, which includes a wand and telemetry interface, and a patient remote control to check battery status and whether the device is on or off. The programmer is used to set up the device, including setup of stimulation and recording, as well as to retrieve data for subsequent review.
  Interventions: Device: Continuous DBS
- Responsive Brain Stimulation (RBS Setting) (Experimental): Eligible participants from Arm 1 will be switch to the RBS intervention.
  Interventions: Device: Responsive Brain Stimulation (RBS Setting)

INTERVENTIONS:
Device: Continuous DBS — The DBS system includes an implantable neurostimulator, CM thalamic leads, and Electrocorticography (ECOG) strips.
  The DBS system will be set to provide continuous stimulation for the 6 months following surgery. Subjects will be seen monthly for evaluation as a part of normal clinical care for DBS. At 6 months, the investigators will determine whether or not the subject is a candidate for responsive brain stimulation (RBS). Qualifying subjects will have the option to have their settings changed in order to participate in the RBS stimulation intervention. Subjects who do not qualify or do not participate will continue to receive this intervention for the duration of the study. These subjects will been seen every 6 months for evaluation as part of normal clinical care for DBS.
  Other Names: Neurostimulator: Medtronic Activa PC+S Device Model 37604; CM thalamic leads: Medtronic Leads Model 3387; ECOG strip leads: The Resume II Medtronic Model 3587A
  Arms: Continuous Deep Brain Stimulation (DBS)
Device: Responsive Brain Stimulation (RBS Setting) — The DBS system includes an implantable neurostimulator, CM thalamic leads, and Electrocorticography (ECOG) strips.
  Six months post-surgery, the DBS system will be set to provide responsive stimulation for the duration of the study. Subjects will be seen every 6 months for evaluation as a part of normal clinical care for DBS.
  Data gathered from the subject during the first 6 months will be used to determine if this intervention is applicable for each individual subject. Subjects who do not qualify will continue to receive the other study intervention.
  Other Names: Neurostimulator: Medtronic Activa PC+S Device Model 37604; CM thalamic leads: Medtronic Leads Model 3387; ECOG strip leads: The Resume II Medtronic Model 3587A
  Arms: Responsive Brain Stimulation (RBS Setting)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of deep brain stimulation (DBS) as a possible new treatment for Tourette Syndrome (TS).

This investigation will (1) test the hypothesis that centromedian (CM) continuous brain stimulation will be an effective, safe method for the treatment of tics in medication refractory TS, (2) will define the intra-operative and post-operative physiological changes, and (3) will test the hypothesis that responsive brain stimulation (RBS) will provide an alternative to chronic DBS in TS.

DETAILED DESCRIPTION:
Normal clinical care for TS includes cognitive behavior therapy, medication, supportive psychotherapy, and/or a combination of the two. To meet entry criteria for this study, you must have already tried these methods and they did not help your symptoms. DBS is considered experimental for the treatment of TS and would not be done as normal clinical care.

Participation in this study will require extensive pre-surgical screening to determine eligibility for DBS surgery, a DBS surgical procedure, and regular follow-ups. Subjects will be seen monthly post surgery for 6 months. After 6 months, data will be assessed and RBS may be offered as a stimulation setting. If so, the stimulator settings will be changed from chronic to responsive. If not, the subject will continue to receive chronic DBS stimulation. Subsequent visits will be scheduled every 6 months until a total of 24 months of study participation.

At the end of the initial 24-month study period, subjects will have the choice of 1) continuing active stimulation at the current setting, 2) continuing stimulation but searching for a new setting, 3) discontinuing stimulation (turning the device off), 4) having the device removed. If the subject continues to receive active stimulation, they will be followed by the PI and seen at yearly intervals until the DBS system is commercially available, FDA approved for the treatment of TS, or unavailable for patient use.

ELIGIBILITY:
Inclusion Criteria:

* Must be 21+ years of age
* Diagnosis of Tourette Syndrome (TS) in accordance to the Diagnostic and Statistical Manual of Mental DIsorders (DSM-V) criteria
* Yale Global Tic Severity Scale (YGTSS) must be ≥35/50 for at least 12 months; Motor Tic subscore must be ≥15
* TS must be causing incapacitation with severe distress, self-injurious behavior, and/or quality of life disruption
* TS must be medication refractory. Criteria to determine if medication refractory is the exact criteria stated by Mink et. al TSA DBS Guidelines published in 2006: Subjects must have been treated by a psychiatrist or neurologist experienced in TS with therapeutic doses of either 1-4 mg/day of haloperidol or 2-8 mg/day of pimozide, risperidone (1-3 mg/day), and aripiprazole (2.5-5 mg/day). Must be at minimum a single trial with an alpha-2 adrenergic agonist (0.1-0.3 mg/day)
* Clinically relevant depression must be pharmacologically treated and deemed stable
* Must have been stabilized for 1 month on TS medication without a dose change prior to surgical intervention. If medication trials resulted in discontinuation of TS medications, the subject must be stabilized for 3 months off TS medicines
* Must be willing to keep TS related medications stable and unchanged throughout the trial
* Must have been offered habit reversal therapy/cognitive behavioral intervention therapy (HRT) if subject did not have it prior to enrollment. (Subjects not required to participate in HRT but it will be highly encouraged, and must be completed prior to start of this study's protocol. Those who improve significantly will be excluded from receiving DBS surgery)
* If tic is focal or addressable by botulinum toxin treatment, the study neurologist will offer to administer a trial of botulinum toxin prior to consideration of surgical therapy. (If the subject chooses not to have the treatment, they cannot participate in the study. If the patient responds satisfactorily and their quality of life significantly improves, they will be excluded)

Exclusion Criteria:

* Any previous neurological intervention including DBS or ablative brain lesions, any metal in the head, and any type of implanted stimulator
* Untreated or unstable anxiety, depression, bipolar disorder, or other Axis I psychiatric disorder
* Presence of psychotic features
* Significant psychosocial factors that can cause increased risk
* The presence of only simple motor tics, a movement disorder other than TS, or medication related movement disorders from TS medications
* Severe medical co-morbidity including cardiovascular disorder, lung disorder, kidney disease, chronic neurological disease, hematological disease, or frailty that impacts tolerability of the surgery as judged by the screening physicians
* Abnormal brain magnetic resonance imaging (MRI) scan, including severe atrophy, hydrocephalus, stroke, structural lesions, demyelinating lesions, or infectious lesions that would potentially confound the outcome or safety of the surgery as judged by the study neurosurgeon
* Dementia or cognitive dysfunction that will place the subject at risk for worsening cognition, and/or may impact the ability to cooperate with tasks involved in the study
* Any attempt or intent of suicide in the last 6 months
* Significant substance abuse or dependence within the last 6 months
* Multiple failed medication treatments of inadequate dose or duration
* History of noncompliance with previous medical and psychosocial treatment efforts
* Severe head banging tics
* Women of child-bearing potential who are pregnant or planning pregnancy (urine pregnancy test required)
* Positive urine drug screen for illicit substances (urine drug screen required)
* History of multiple surgical procedures with poor outcomes
* Unexplained gaps in medical history
* Pending lawsuits or other legal action

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Okun, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Cagle JN, Okun MS, Cernera S, Eisinger RS, Opri E, Bowers D, Ward H, Foote KD, Gunduz A. Embedded Human Closed-Loop Deep Brain Stimulation for Tourette Syndrome: A Nonrandomized Controlled Trial. JAMA Neurol. 2022 Oct 1;79(10):1064-1068. doi: 10.1001/jamaneurol.2022.2741. PMID 36094652
- See also: UF Center for Movement Disorders & Neurorestoration — http://movementdisorders.ufhealth.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from 3/20/14 to 3/16/20. Some participants were referrals from other centers and some were from the UF Health Neurology clinic.
Groups:
- First Period: Continuous DBS; Second Period: Switch to Responsive DBS in Qualified Patients: The surgical intervention requires implantation of a DBS system: one CM thalamic leads per hemisphere, one Electrocorticography (ECOG) strip per hemisphere, and two neurostimulators implanted in the chest. The strip provides an interface for brain activity to be monitored.
  The system includes a programmer with a telemetry interface and a patient remote to check battery and device status. The programmer is used to set up the device, i.e., stimulation and recording, and retrieve data for subsequent review.
  First Period: The system will be set to provide continuous deep brain stimulation (CDBS) for the 6 months postsurgery. Subjects will be evaluated monthly as part of normal clinical care for DBS.
  Second Period: At 6 months, the investigators will determine whether a subject is a candidate for responsive brain stimulation (RBS). A neuromarker that detects tics significantly must be identified for a subject to receive the second intervention. Qualifying subjects will have the option to change their settings to participate in the RBS stimulation intervention. Subjects who do not qualify or do not participate will continue to receive this intervention for the duration of the study. Subjects will been seen every 6 months for evaluation as part of normal clinical care for DBS.
Period: Continuous DBS
Arm/Group | First Period: Continuous DBS; Second Period: Switch to Responsive DBS in Qualified Patients
Started | 10
Qualify for Second Intervention at the End of First Intervention | 10
Completed | 10
Not Completed | 0
Period: Responsive DBS
Arm/Group | First Period: Continuous DBS; Second Period: Switch to Responsive DBS in Qualified Patients
Started | 8 (2 participants' study period finished before firmware update was available for the second period.)
Completed | 5
Not Completed | 3
Not completed — CDBS parameters of 3 subjects | 3

BASELINE CHARACTERISTICS:
Population: Patients with Tourette Syndrome that have been deemed candidates for deep brain stimulation (DBS) surgery.
Groups:
- Deep Brain Stimulation (DBS): The surgical intervention requires implantation of a DBS system: one CM thalamic leads per hemisphere, one Electrocorticography (ECOG) strip per hemisphere, and two neurostimulators implanted in the chest. The strip provides an interface for brain activity to be monitored.
  The system includes a programmer with a telemetry interface, and a patient remote to check battery and device status. The programmer is used to set up the device, i.e., stimulation and recording, and retrieve data for subsequent review.
  The system will be set to provide continuous stimulation for the 6 months postsurgery. Subjects will be seen monthly for evaluation as a part of normal clinical care for DBS. At 6 months, the investigators will determine whether a subject is a candidate for responsive brain stimulation (RBS). Qualifying subjects will have the option to have their settings changed in order to participate in the RBS stimulation intervention. Subjects who do not qualify or do not participate will continue to receive this intervention for the duration of the study. Subjects will been seen every 6 months for evaluation as part of normal clinical care for DBS.
Arm/Group | Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Yale Global Tic Severity Scale (YGTSS) [Mean (Full Range); unit: units on the YGTSS scale] — YGTSS is a questionnaire that has a range of 0-50, with higher values corresponding to more severe symptoms. The goal of the interventions is to decrease the presurgical baseline measure.
  units on the YGTSS scale | 39 [0 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 40% Reduction in Total Tics on the Yale Global Tic Severity Scale (YGTSS) With CDBS (Period 1)
Description: The Yale Global Tic Severity Scale (YGTSS) is a 10-item semi-structured clinician-rating instrument that provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic symptoms. The items pertaining to the tic ratings are scored on two subscales: motor tics and phonic tics. Behaviors are rated on a 6-point scale. The total scale has been used in this study and has a range of 0-50. A higher score indicates a higher severity of symptoms.
  Patients reach the outcome measure with a 40% reduction of YGTSS at month 6 post-op compared to baseline (i.e., 40% improvement in their tic severity scale).
Time Frame: Baseline to 6 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 10
Participants | 4
Statistical Analysis 1: Comparison: Deep Brain Stimulation (DBS); At 6 months post-surgery the YGTSS scores of each subjects is statistically tested against their baseline scores. A decrease in this tic severity scale means that the severity of the tics have reduced. Hence, we performed a superiority test, which statistically verifies if the reduction in the tic severity scale was meaningful; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .3

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Continuous Deep Brain Stimulation (DBS): Subjects' DBS surgical intervention requires implantation of two bilateral DBS system: a CM thalamic lead,an ECOG strip leads, one neurostimulator implanted in the chest per hemisphere.
  Neurostimulator and leads system includes a programmer with a telemetry interface, and a patient remote control to check device status. The programmer is used to set up the stimulation and signal recording to retrieve data for subsequent review.
  The DBS system will provide continuous stimulation for the 6 months following surgery. Subjects will be seen monthly for evaluation as a part of normal clinical care for DBS. At 6 months, the investigators will determine whether the subject is a candidate for responsive brain stimulation (RBS). Qualifying subjects will have the option to have their settings changed in order to participate in the RBS stimulation intervention. Subjects who do not qualify or do not participate will continue to receive this intervention for the duration of the study.
  Six months post-surgery, the DBS system will be set to provide responsive stimulation for the duration of the study. Subjects will be seen every 6 months for evaluation as a part of normal clinical care for DBS.
  Data gathered from the subject during the first 6 months will be used to determine if this intervention is applicable for each individual subject. Subjects who do not qualify will continue to receive the other study intervention.
- Responsive Brain Stimulation (RBS): At 6 months, the investigators will determine whether the subject is a candidate for responsive brain stimulation (RBS). Qualifying subjects will have the option to have their settings changed in order to participate in the RBS stimulation intervention. Subjects who do not qualify or do not participate will continue to receive this intervention for the duration of the study.
Arm/Group | Continuous Deep Brain Stimulation (DBS) | Responsive Brain Stimulation (RBS)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/5
Other Adverse Events (participants affected / at risk) | 10/10 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Deep Brain Stimulation (DBS) (N=10) | Responsive Brain Stimulation (RBS) (N=5)
renal and urinary disorder, other (Renal and urinary disorders) | 1 (1) | NA — bladder prolapse
esophageal ulcers (Gastrointestinal disorders) | 1 (1) | NA
rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | NA
rectal pain (Gastrointestinal disorders) | 1 (1) | NA — rectal prolapse
gastric ulcer (Gastrointestinal disorders) | 1 (1) | NA
pelvic pain (Reproductive system and breast disorders) | 1 (1) | NA — uterine prolapse
psychiatric disorders - other, mood disorder (Psychiatric disorders) | 1 (2) | NA — psychiatric inpatient hospitalization
injury, poisoning and procedural complications, other - concussion (Injury, poisoning and procedural complications) | 1 (1) | NA — concussion from a car accident
psychosis (Psychiatric disorders) | 1 (1) | NA
device related infection (Infections and infestations) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Deep Brain Stimulation (DBS) (N=10) | Responsive Brain Stimulation (RBS) (N=5)
akathisia (Nervous system disorders) | 2 (2) | NA
allergic reaction (Immune system disorders) | 1 (1) | NA
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
anxiety (Psychiatric disorders) | 4 (5) | NA
cholecystitis (Hepatobiliary disorders) | 1 (1) | NA — gall bladder inflammation
dehydration (Metabolism and nutrition disorders) | 1 (1) | NA
depression (Psychiatric disorders) | 3 (3) | NA
dysarthria (Nervous system disorders) | 1 (1) | NA
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
fatique (General disorders) | 1 (1) | NA
flushing (Vascular disorders) | 1 (1) | NA
gastroenteritis (Gastrointestinal disorders) | 1 (1) | NA
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | NA
gastrointestinal, other - excessive salivation (Gastrointestinal disorders) | 1 (1) | NA
headache (Nervous system disorders) | 7 (13) | NA
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
insomnia (Psychiatric disorders) | 2 (2) | NA
irregular menstruation (Reproductive system and breast disorders) | 1 (2) | NA
joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
localized edema (General disorders) | 4 (8) | NA
mania (Psychiatric disorders) | 1 (1) | NA — hypomania
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | NA — myalgia - hip
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | NA
nausea (Gastrointestinal disorders) | 4 (7) | NA
neck pain (Musculoskeletal and connective tissue disorders) | 1 (5) | NA
neoplasms benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA — ovarian cysts
neuralgia (Nervous system disorders) | 1 (1) | NA
pain (General disorders) | 2 (3) | NA — pain at IPG
parasthesia (Nervous system disorders) | 3 (7) | NA
psychiatric disorders - other, nightmares (Psychiatric disorders) | 1 (1) | NA
psychiatric disorders, other - tics (Psychiatric disorders) | 3 (5) | NA
psychiatric disorders, other - pseudobulbar affect (Psychiatric disorders) | 1 (1) | NA
psychosis (Psychiatric disorders) | 1 (1) | NA
rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | NA
rash maculo-papular with pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | NA
scalp pain (Skin and subcutaneous tissue disorders) | 3 (3) | NA
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — sinus cavities blocked - surgically cleared
sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
skin infection (Skin and subcutaneous tissue disorders) | 1 (4) | NA
spasticity (Nervous system disorders) | 1 (1) | NA
suicidal ideation (Psychiatric disorders) | 1 (2) | NA
thrush (Infections and infestations) | 1 (1) | NA
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | NA
vomiting (Gastrointestinal disorders) | 5 (7) | NA
weight gain (Investigations) | 1 (1) | NA
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT02056873/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT02056873/ICF_001.pdf